CLINICAL TRIAL: NCT06058572
Title: Randomized Trial to Study the Effect of Rifaximin on Gut Microbiome Diversity Post Allogeneic Stem Cell Transplant in Acute Leukemia.
Brief Title: Effect of Rifaximin on Gut Bacterial Flora Post Stem Cell Transplant in Patients With Acute Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 900872
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Acute Leukemia
Keywords: Rifaximin; Gut Microbiome
MeSH Terms: interventions — Rifaximin

STUDY DESIGN:
Intervention Model Description: Interventional Arm : Tab Rifaximin 200 mg along with allogeneic stem cell transplant
  Standard Arm : Allogeneic stem cell transplant alone (with no anti-microbial prophylaxis)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rifaxmin +aHSCT (Experimental): drug rifaximin 200 mg tablet form orally twice daily (with or without food) from day-8 of transplant to day + 60 of transplant
  Interventions: Drug: Rifaximin 200Mg Tab
- aHSCT alone (Active Comparator): control arm will underwent allogenic hematopoietic stem cell transplantation procedure as per standard of care
  Interventions: Procedure: allogenic hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: Rifaximin 200Mg Tab — Drug rifaximin 200 mg tablet form orally twice daily (with or without food) from day-8 of transplant to day + 60 of transplant
  Arms: Rifaxmin +aHSCT
Procedure: allogenic hematopoietic stem cell transplantation — Control arm will undergo allogenic hematopoietic stem cell transplantation as standard of care
  Arms: aHSCT alone

SUMMARY:
* Goal: This study is a randomized phase II interventional study. The purpose of this study is to see if addition of oral rifaximin tablets during allogeneic stem cell transplant can improve the quality of gut microbiome and reduce chances of death, infections and graft versus host disease (GVHD) post-transplant.
* The study objectives are as follows:
* Primary Objective: To determine the impact of rifaximin on gut microbial diversity and compare it with controls.
* Secondary Objectives: a. To determine non-relapse mortality at 1-year post transplant in patients who receive peri-transplant transplant rifaximin and compare it with controls.
* b. To compare the incidence of severe GVHD in patients who receive peri-transplant rifaximin with the controls.
* c. To determine impact of gut decontamination with rifaximin on incidence of MDR sepsis and usage of higher antibiotics (e.g. Carbapenems, colistin, tigecycline, ceftazidime avibactum and ceftriaxone-sulbactam EDTA) in first 6 months post BMT.
* d. To determine the impact of rifaximin induced gut manipulation on immune reconstitution, T cell repertoire post-transplant and cytokine profile.
* Exploratory objective: To use single cell transcriptomics (SCT) to identify immune cell profile in gut biopsies post allogeneic stem cell transplant whenever biopsy is done, to correlate the impact of microbiome on gut immunity.
* Intervention: Tab Rifaximin 200 mg will be given orally twice daily from day -8 to day +60 of allogeneic stem cell transplant in acute leukemia patients. This will be in addition to standard of care post-transplant treatment.
* Comparator Agent: Standard of care treatment including standard anti GVHD measures, antibiotic support and transfusions as needed.

DETAILED DESCRIPTION:
The gut microbiome plays a significant role in modulating the immune re-constitution post allogeneic stem cell transplant (ASCT). Low gut microbial diversity has been consistently associated with poor outcomes of transplant including increased incidence of acute graft versus host disease (aGVHD), post-transplant bacterial sepsis and non-relapse mortality (NRM). However, the exact mechanism by which gut microbiome influences local as well as systemic immunity is not completely known, and is thought to be due to the impact of microbial metabolites on intestinal epithelial cells and host antigen-presenting cells. Understanding these mechanisms and modulating the microbiome may be crucial to improving transplant outcomes. Rifaximin is a locally acting antibiotic that has been approved for manipulating the gut microbiome in hepatic failure. It is unique because of its ability to clear pathogenic bacteria, while preserving the anaerobic commensals. It can potentially modify the gut microbiome to increase the alpha diversity and this may help reduce aGVHD, infectious complications, and mortality post-transplant. High incidence of multidrug resistant sepsis and frequent use of broad spectrum antibiotics in India, would result in higher rates of dysbiotic gut- making microbiome manipulation to improve transplant outcomes more relevant in our country. We are proposing a randomized controlled trial to understand the benefits of modulating the gut microbiome in patients of ASCT while investigating the local and global immune repertoire using single cell sequencing and multicolour flow cytometry.

Study design: Single center, open-labeled, phase II study, randomized controlled trial.

Primary Objective: To determine the impact of rifaximin on gut microbial alpha diversity and compare it with controls.

Secondary Objectives:

To determine impact of rifaximin on 1 year non relapse mortality post-transplant, incidence of grade III/IV aGVHD, incidence of MDR sepsis, patterns of immune cell reconstitution, and cytokine profile post-transplant.

Exploratory objective: To use single-cell transcriptomics (SCT) to identify immune cell profiles in gut biopsies post ASCT in order to get insights into the impact of the microbiome on local gut immunity.

Study population: Adult patients who undergo ASCT at the Tata Memorial Centre.

Study Methodology in brief: Patients would be randomized to receive either oral tablet rifaximin 200 mg twice daily along with standard posttransplant treatment or to receive standard of care treatment alone. Stool samples and blood samples will be collected at different time points for microbiome analysis and immune cell profiling respectively. We plan to perform 16s rRNA-based next-generation sequencing of all variable regions using a phased primer approach using stool DNA as a template. Gut microbiome diversity will be calculated using the inverse Simpson index. Immune cell profile would be analyzed using 16 color flow cytometry. In selected cases where patients undergo colonoscopic gut biopsy for aGVHD, we will also obtain samples for transcriptome sequencing. This will help us understand how immune cells interact with gut mucosa and microbiome in patients of aGVHD

ELIGIBILITY:
Inclusion Criteria:

* Adults with acute leukemia undergoing allogeneic stem cell transplant.
* ECOG performance status 0, 1 or 2.
* Adequate Liver function

Exclusion Criteria:

* Known hypersensitivity to rifaximin or other rifampicin antimicrobial agents
* Current or past history of inflammatory bowel disease
* History of major bowel resection or presence of colostomy.
* Ongoing Verapamil, ketoconazole or itraconazole.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2027-08-02 (Estimated); Study Completion 2027-08-02 (Estimated)

PRIMARY OUTCOMES:
Impact of rifaximin on gut microbial diversity. | 14 days post transplant
  Gut microbial diversity as measured by inverse Simpson index (ISI) on stool samples on day 14 post transplant in Rifaximin arm and in controls.

SECONDARY OUTCOMES:
Non relapse mortality | 1 year post transplant
  Non relapse mortality (NRM) at 1 year post transplant in patients who receive peri-transplant transplant rifaximin and in controls
Incidence of severe (grade III/IV) acute graft versus host disease | 1 year post transplant
  Incidence of severe (grade III/IV) acute graft versus host disease (aGVHD) in patients who receive peri-transplant rifaximin and in control arm.
Impact of gut decontamination with rifaximin on incidence of multidrug resistant sepsis post transplant. | 6 months post transplant
  Incidence of multidrug resistant (MDR) sepsis and usage of higher antibiotics (e.g. Carbapenems, colistin, tigecycline, ceftazidime avibactam and ceftriaxone-sulbactam EDTA) in first 6 months post BMT in both rifaximin arm and in controls.
Impact of rifaximin induced gut manipulation on immune reconstitution | 1 year post transplant
  Immune-reconstitution, T cell repertoire post transplant as measured by multicolor flow-cytometry in patients who receive rifaximin and in controls.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Anant Gokarn, Gokarn, Principal Investigator — Advanced Centre for Treatment, Research and Education in Cancer
Locations (1):
- Actrec Tmc, Navi Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No
No not shared